CLINICAL TRIAL: NCT03537196
Title: Towards HCV Elimination: Evaluation of an Integrated Model of HCV Care Targeting People Who Inject Drugs in Hai Phong, Vietnam
Brief Title: DRug Use & Infections in ViEtnam - Hepatitis C (DRIVE-C)
Acronym: DRIVE-C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12380 DRIVE-C
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Hepatitis C; Drug Use; Viral Hepatitis C
Keywords: People who inject drugs; Hepatitis C; Direct Acting Antiviral; HCV Elimination; Vietnam; Viral hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; daclatasvir; Ribavirin

STUDY DESIGN:
Intervention Model Description: All patients with detectable HCV RNA, eligible for treatment, will receive Direct Acting Antiviral drugs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- All patients (Other): All patients will receive sofosbuvir 400-mg and daclatasvir 60-mg (1 tablet each per day) during 12 weeks.
  Interventions: Drug: Sofosbuvir 400 mg and Daclatasvir 60 mg
- HIV/HCV co-infected patients (Other): For HIV/HCV co-infected patients receiving efavirenz or nevirapine, daclatasvir dose will be increased to 90-mg per day (sofosbuvir 400 mg and daclatasvir 90 mg)
  Interventions: Drug: Sofosbuvir 400 mg and Daclatasvir 90 mg
- Cirrhosis (Other): In case of cirrhosis : ribavirin will be added to sofosbuvir / daclatasvir 12 weeks
  Interventions: Drug: Ribavirin
- Cirrhosis with ribavirin contra-indication (Other): In case of cirrhosis with ribavirin contra-indication : sofosbuvir and daclatasvir for 24 weeks
  Interventions: Drug: Sofosbuvir and Daclatasvir for 24 weeks

INTERVENTIONS:
Drug: Sofosbuvir 400 mg and Daclatasvir 60 mg — All patients will receive sofosbuvir 400-mg and daclatasvir 60-mg (1 tablet each per day) during 12 weeks.
  Arms: All patients
Drug: Sofosbuvir 400 mg and Daclatasvir 90 mg — For HIV/HCV co-infected patients receiving efavirenz or nevirapine, daclatasvir dose will be increased to 90-mg per day.
  Arms: HIV/HCV co-infected patients
Drug: Ribavirin — In case of cirrhosis:
  * Ribavirin will be added to sofosbuvir/daclatasvir during the 12 weeks of treatment. The dose will be adapted to the patient weight although the vast majority of patients (weight < 75 kg) will receive 500 mg x 2/day.
  * In case of ribavirin contra-indication or side effects leading to ribavirin discontinuation, sofosbuvir/daclatasvir will be used 24 weeks.
  Arms: Cirrhosis
Drug: Sofosbuvir and Daclatasvir for 24 weeks — In case of cirrhose and of ribavirin contra-indication or side effects leading to ribavirin discontinuation, sofosbuvir/daclatasvir will be used 24 weeks.
  Arms: Cirrhosis with ribavirin contra-indication

SUMMARY:
The study aims to assess the effectiveness of a model of hepatitis C screening and integrated care, targeting people who inject drugs (PWIDs) in Hai Phong, Vietnam. In a wider perspective, this model linked to mass screening through repeated Respondent Driven Sampling (RDS) surveys, to simplified treatment protocol, and to large community-based support to improve referral to care, retention in care, adherence to treatment and prevention of reinfection, may have the potential to eliminate HCV among PWIDs in this city.

DETAILED DESCRIPTION:
Objectives :

The primary objective of this study is to assess the effectiveness of a model of hepatitis C screening and integrated care targeting PWIDs in Hai Phong, Vietnam.

This model will encompass all steps involved in achieving HCV cure among PWIDs:

i) Mass detection of hepatitis C infection among PWIDs: in the community through a large community-based Respondent Driven Sampling survey (RDS); and in HIV out-patient clinics and methadone treatment centers where serological testing should have been made, but not HCV RNA to confirm hepatitis C infection.

ii) a community-based support to improve referral to specific care for those with hepatitis C infection; iii) a HCV care system delivery integrated within the existing health system with a simplified treatment protocol taking into account PWIDs specificities such as frequent HIV co-infection and methadone treatment; iv) an optimized treatment adherence through a combination of health care therapeutic education and CBO support; v) an increase in harm reduction activities to encompass HCV risk transmission and to prevent HCV reinfection.

Secondary objectives are:

* to assess all steps of the hepatitis C cascade of care (Hepatitis C infection diagnosis; HCV care enrolment; HCV treatment initiation; HCV treatment success);
* to assess the occurrence of adverse events (death, morbidity) and drug-related side-effects;
* to evaluate adherence to HCV treatment;
* to determine factors associated with treatment failure defined by a positive HCV RNA 12 weeks after the end of HCV treatment;
* to estimate the reinfection rate at the end of the study and to identify risk factors of HCV reinfection;
* to project the impact and cost-effectiveness of the implemented HCV treatment intervention.

Study design : the effectiveness-implementation hybrid study type 1 design will simultaneously allow assessing the effectiveness of Direct-Acting Antivirals (DAA) care strategy among PWIDs in Vietnam, and the potential obstacles to widespread implementation.

The strategy of care includes a large community-based mass screening, a simplified treatment protocol based on a combination of DAAs, taking into account co-morbidities (addiction, HIV), physician training and important support of Community Based Organizations (CBO's) for linkage to care after screening, treatment adherence and prevention of reinfection after cure.

In addition, 2 others components are included in the study:

* A modeling exercise to assess the impact of the intervention at the population level,
* A cost-effectiveness analysis to further inform policy-makers.

Patients will be followed for 48 weeks after initiating HCV treatment. The estimated enrolment is 1050 participants.

Study population: people who currently inject drugs or who have recently started opioid substitution treatment.

Implementation: The study is linked to the NIDA RO1 DA041978 / ANRS 12353 DRIVE project. Participant recruitment will take place through DRIVE RDS survey and DRIVE cohort follow-up visit in two community sites managed by peer-groups in Hai Phong. All participants with positive HCV serology will be screened for hepatitis C and positive HCV RNA will be proposed for DAA treatment in 3 hospital-based HCV clinics. All participants will attend 9 study visits, comprising of clinical examination, blood collection for side effects and viral load assessment, therapeutic education, questionnaires on alcohol use, on sexual, drug use and other behaviors focusing on HCV infection risks or HCV reinfection risks and on quality of life, and harm reduction activities with the support of CBOs.

ELIGIBILITY:
INCLUSION CRITERIA

* Participants of the ANRS 12353/NIDA ROI DA 041978 DRIVE study (age > 18 years; positive urine test for heroin an/o methamphetamine & skin marks of injection ) who either participated to the DRIVE RDS3 survey, or to the HIV-positive and HIV-negative DRIVE cohorts;
* Hepatitis C infection defined by a positive HCV RNA
* Signed informed consent form

EXCLUSION CRITERIA

* Severe associated diseases requiring specific treatment (including all specific AIDS defining illnesses, any severe sepsis, severe decompensated cirrhosis, suspicion of hepatocellular carcinoma);
* Any condition which might, in the investigator's opinion, compromise the safety of the patient by participating in the study including very severe clinical condition;
* Previous history of DAA use;
* Contraindication for treatment with sofosbuvir or daclatasvir;
* For women of childbearing potential i.e. women of childbearing age who are not menopausal, or permanently sterilized or not refraining from sexual activity:
* Pregnancy and breastfeeding
* Refusal to use a contraceptive method
* Renal failure with creatinine clearance ≤ 30 milliliter per minute;
* Person deprived of freedom by a judicial or administrative decision;
* Person who plan to move out from Hai Phong in the next 12 months;
* Person unable to understand the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of all patients in success of the model of care | Week 48
  Proportion of patients with HCV RNA < 15 IU/mL at the end of the study among patients who have signed the informed consent.

SECONDARY OUTCOMES:
Proportion of patients with detectable HCV RNA | Screening pre-inclusion
  Proportion of patients with HCV RNA > 15 IU/mL among those with positive HCV Ab
Proportion of patients enrolled in care | Pre-inclusion visit
  Proportion of patients with HCV RNA > 15 IU/mL who attended the pre inclusion visit at HCV clinic among those with hepatitis C infection;
Proportion of patients initiating DAA treatment | Initiation treatment visit
  Proportion of patients who initiate the treatment among patients enrolled in care and eligible for treatment
Proportion of patients cured | Week 24
  Number of patients with HCV RNA < 15 IU/mL among those initiating the treatment eligible
Rate of reinfection | Week 48
  Number of patients with HCV RNA ≥ 15 IU/mL at the end of the study among cured patients
Rate of mortality | Week 48
  Rate of deaths among all participants with hepatitis C infection
Frequency, type and time to grade 3 or 4 adverse clinical or biological events. | Week 48
  All adverse events will be graded according to the ANRS adverse events grading table
Frequency, type and time to drug-related clinical or biological adverse reactions | Week 48
  All drug-related clinical or biological adverse reactions of grade 3 or 4 or leading to treatment interruption
Adherence assessment | Week 12
  Self-questionnaire on DAA drug intake and drug accountability for DAA
Factors associated with HCV treatment failure | Week 24
  Socio-demographic, co-infection, virological, adherence, behavioral, psychiatric disorders, intervention contact, recent incarceration, homelessness factors
Factors associated with HCV reinfection | Week 48
  Socio-demographic, co-infection, virological, adherence, behavioral, psychiatric disorders, intervention contact, recent incarceration, homelessness factors
Effect of the HCV treatment intervention | Week 48
  Estimation of the impact of the intervention on HCV infections and DALYs averted, QALYs saved, HCV incidence and prevalence as projected by the model under various scenarios
Incremental cost-effectiveness ratio (ICER) | Week 48
  Estimation of the mean ICER which will be compared against standard thresholds for intervention's being cost-effective in LMIC settings

CONTACTS AND LOCATIONS:
Overall Officials: KHUE M. PHAM, MD, PhD, Principal Investigator — Hai Phong University of Medicine and Pharmacy, Vietnam; DIDIER LAUREILLARD, MD, Principal Investigator — Nîmes University Hospital, France; NICOLAS NAGOT, MD, PhD, Study Director — Pathogenesis and Control of Chronic Infections (PCCI) UMR 1058 - INSERM, Univ Montpellier, EFS, Montpellier, France
Locations (2):
- Vietnam (2):
  - Hai Phong University of Medicine and Pharmacy, Haiphong
  - Viet Tiep Hospital, Haiphong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gower E, Estes C, Blach S, Razavi-Shearer K, Razavi H. Global epidemiology and genotype distribution of the hepatitis C virus infection. J Hepatol. 2014 Nov;61(1 Suppl):S45-57. doi: 10.1016/j.jhep.2014.07.027. Epub 2014 Jul 30. PMID 25086286
- [Background] Mohd Hanafiah K, Groeger J, Flaxman AD, Wiersma ST. Global epidemiology of hepatitis C virus infection: new estimates of age-specific antibody to HCV seroprevalence. Hepatology. 2013 Apr;57(4):1333-42. doi: 10.1002/hep.26141. Epub 2013 Feb 4. PMID 23172780
- [Background] Sereno L, Mesquita F, Kato M, Jacka D, Nguyen TT, Nguyen TN. Epidemiology, responses, and way forward: the silent epidemic of viral hepatitis and HIV coinfection in Vietnam. J Int Assoc Physicians AIDS Care (Chic). 2012 Sep-Oct;11(5):311-20. doi: 10.1177/1545109712453939. Epub 2012 Jul 24. PMID 22828983
- [Background] Clatts MC, Colon-Lopez V, Giang LM, Goldsamt LA. Prevalence and incidence of HCV infection among Vietnam heroin users with recent onset of injection. J Urban Health. 2010 Mar;87(2):278-291. doi: 10.1007/s11524-009-9417-9. PMID 20041309
- [Background] Gish RG, Bui TD, Nguyen CT, Nguyen DT, Tran HV, Tran DM, Trinh HN; International Group for Liver Health in Viet Nam. Liver disease in Viet Nam: screening, surveillance, management and education: a 5-year plan and call to action. J Gastroenterol Hepatol. 2012 Feb;27(2):238-47. doi: 10.1111/j.1440-1746.2011.06974.x. PMID 22098550
- [Background] Kallman JB, Tran S, Arsalla A, Haddad D, Stepanova M, Fang Y, Wrobel VJ, Srishord M, Younossi ZM. Vietnamese community screening for hepatitis B virus and hepatitis C virus. J Viral Hepat. 2011 Jan;18(1):70-6. doi: 10.1111/j.1365-2893.2010.01278.x. PMID 20196807
- [Background] Pham DA, Leuangwutiwong P, Jittmittraphap A, Luplertlop N, Bach HK, Akkarathamrongsin S, Theamboonlers A, Poovorawan Y. High prevalence of Hepatitis C virus genotype 6 in Vietnam. Asian Pac J Allergy Immunol. 2009 Jun-Sep;27(2-3):153-60. PMID 19839502
- [Background] Tanimoto T, Nguyen HC, Ishizaki A, Chung PT, Hoang TT, Nguyen VT, Kageyama S, Oka S, Pham VT, Ichimura H. Multiple routes of hepatitis C virus transmission among injection drug users in Hai Phong, Northern Vietnam. J Med Virol. 2010 Aug;82(8):1355-63. doi: 10.1002/jmv.21787. PMID 20572071
- [Background] Liang TJ, Ghany MG. Current and future therapies for hepatitis C virus infection. N Engl J Med. 2013 May 16;368(20):1907-17. doi: 10.1056/NEJMra1213651. PMID 23675659
- [Background] Pawlotsky JM, Feld JJ, Zeuzem S, Hoofnagle JH. From non-A, non-B hepatitis to hepatitis C virus cure. J Hepatol. 2015 Apr;62(1 Suppl):S87-99. doi: 10.1016/j.jhep.2015.02.006. PMID 25920094
- [Background] Martin NK, Vickerman P, Grebely J, Hellard M, Hutchinson SJ, Lima VD, Foster GR, Dillon JF, Goldberg DJ, Dore GJ, Hickman M. Hepatitis C virus treatment for prevention among people who inject drugs: Modeling treatment scale-up in the age of direct-acting antivirals. Hepatology. 2013 Nov;58(5):1598-609. doi: 10.1002/hep.26431. Epub 2013 Aug 26. PMID 23553643
- [Background] Grebely J, Matthews GV, Lloyd AR, Dore GJ. Elimination of hepatitis C virus infection among people who inject drugs through treatment as prevention: feasibility and future requirements. Clin Infect Dis. 2013 Oct;57(7):1014-20. doi: 10.1093/cid/cit377. Epub 2013 May 31. PMID 23728143
- [Background] European Association for the Study of the Liver. EASL Recommendations on Treatment of Hepatitis C 2016. J Hepatol. 2017 Jan;66(1):153-194. doi: 10.1016/j.jhep.2016.09.001. Epub 2016 Sep 22. No abstract available. PMID 27667367
- [Background] Bruggmann P, Grebely J. Prevention, treatment and care of hepatitis C virus infection among people who inject drugs. Int J Drug Policy. 2015 Feb;26 Suppl 1:S22-6. doi: 10.1016/j.drugpo.2014.08.014. Epub 2014 Aug 30. PMID 25245939
- [Background] Des Jarlais D, Duong HT, Pham Minh K, Khuat OH, Nham TT, Arasteh K, Feelemyer J, Heckathorn DD, Peries M, Moles JP, Laureillard D, Nagot N; (The Drive Study Team). Integrated respondent-driven sampling and peer support for persons who inject drugs in Haiphong, Vietnam: a case study with implications for interventions. AIDS Care. 2016 Oct;28(10):1312-5. doi: 10.1080/09540121.2016.1178698. Epub 2016 May 13. PMID 27178119
- [Background] Guidelines for the Screening Care and Treatment of Persons with Chronic Hepatitis C Infection: Updated Version. Geneva: World Health Organization; 2016 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK362924/ PMID 27227200
- [Background] Nguyen Truong T, Laureillard D, Lacombe K, Duong Thi H, Pham Thi Hanh P, Truong Thi Xuan L, Chu Thi N, Luong Que A, Vu Hai V, Nagot N, Tuaillon E, Dominguez S, Lemoine M. High Proportion of HIV-HCV Coinfected Patients with Advanced Liver Fibrosis Requiring Hepatitis C Treatment in Haiphong, Northern Vietnam (ANRS 12262). PLoS One. 2016 May 5;11(5):e0153744. doi: 10.1371/journal.pone.0153744. eCollection 2016. PMID 27148964
- [Background] Martin NK, Hickman M, Hutchinson SJ, Goldberg DJ, Vickerman P. Combination interventions to prevent HCV transmission among people who inject drugs: modeling the impact of antiviral treatment, needle and syringe programs, and opiate substitution therapy. Clin Infect Dis. 2013 Aug;57 Suppl 2(Suppl 2):S39-45. doi: 10.1093/cid/cit296. PMID 23884064
- [Background] Altice FL, Azbel L, Stone J, Brooks-Pollock E, Smyrnov P, Dvoriak S, Taxman FS, El-Bassel N, Martin NK, Booth R, Stover H, Dolan K, Vickerman P. The perfect storm: incarceration and the high-risk environment perpetuating transmission of HIV, hepatitis C virus, and tuberculosis in Eastern Europe and Central Asia. Lancet. 2016 Sep 17;388(10050):1228-48. doi: 10.1016/S0140-6736(16)30856-X. Epub 2016 Jul 14. PMID 27427455
- [Background] Vickerman P, Martin N, Turner K, Hickman M. Can needle and syringe programmes and opiate substitution therapy achieve substantial reductions in hepatitis C virus prevalence? Model projections for different epidemic settings. Addiction. 2012 Nov;107(11):1984-95. doi: 10.1111/j.1360-0443.2012.03932.x. Epub 2012 Jul 12. PMID 22564041
- [Background] Smith DJ, Combellick J, Jordan AE, Hagan H. Hepatitis C virus (HCV) disease progression in people who inject drugs (PWID): A systematic review and meta-analysis. Int J Drug Policy. 2015 Oct;26(10):911-21. doi: 10.1016/j.drugpo.2015.07.004. Epub 2015 Jul 26. PMID 26298331
- [Background] Conti F, Buonfiglioli F, Scuteri A, Crespi C, Bolondi L, Caraceni P, Foschi FG, Lenzi M, Mazzella G, Verucchi G, Andreone P, Brillanti S. Early occurrence and recurrence of hepatocellular carcinoma in HCV-related cirrhosis treated with direct-acting antivirals. J Hepatol. 2016 Oct;65(4):727-733. doi: 10.1016/j.jhep.2016.06.015. Epub 2016 Jun 24. PMID 27349488
- [Derived] Laureillard D, Binh NT, Vinh VH, Hong TT, Quillet C, Thanh NTT, Vallo R, Quynh BTN, Moles JP, Oanh KTH, Huong DT, Rapoud D, Feelemyer J, Michel L, Vickerman P, Fraser H, Weiss L, Lemoine M, Lacombe K, Jarlais DD, Khue PM, Nagot N. High Efficiency and Safety of Hepatitis C Treatment Among People Who Inject Drugs in Vietnam. J Viral Hepat. 2025 Nov;32(11):e70090. doi: 10.1111/jvh.70090. PMID 41017776
- [Derived] Rapoud D, Quillet C, Pham Minh K, Vu Hai V, Nguyen Thanh B, Nham Thi Tuyet T, Tran Thi H, Moles JP, Vallo R, Michel L, Feelemyer J, Weiss L, Lemoine M, Vickerman P, Fraser H, Duong Thi H, Khuat Thi Hai O, Des Jarlais D, Nagot N, Laureillard D; DRIVE-C Study Group. Towards HCV elimination among people who inject drugs in Hai Phong, Vietnam: study protocol for an effectiveness-implementation trial evaluating an integrated model of HCV care (DRIVE-C: DRug use & Infections in ViEtnam-hepatitis C). BMJ Open. 2020 Nov 18;10(11):e039234. doi: 10.1136/bmjopen-2020-039234. PMID 33208326